CLINICAL TRIAL: NCT06508385
Title: The Effect of Perception of Improvement Provided Virtual Reality Environment on Symptom Presence and Severity in Patients With Fibromyalgia
Brief Title: The Effect of Perception of Improvement in Patients With Fibromyalgia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Nilufer Kablan, Assoc. prof, Istanbul Medeniyet University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023/0689
Record Dates: First submitted 2024-07-12; First posted 2024-07-18 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Fibromyalgia
Keywords: functional brain activity; Pain; Tissue properties
MeSH Terms: conditions — Fibromyalgia; Pain | interventions — Breathing Exercises

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Double
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (Active Comparator): NLP-supported patient education will be given and breath therapy will be applied to the Control Group
  Interventions: Other: Breathing exercise
- Virtual Reality Group-1 (Experimental): NLP-supported patient education will be given. Visual feedback and metaphor-assisted breathing therapy over the three most painful points in the McGill-Melzack Pain Scale (real painful points) were given to this group in virtual reality environment.
  Interventions: Other: Breathing exercise
- Virtual Reality Group-2 (Experimental): NLP-supported patient education will be given. Visual feedback and metaphor-assisted breathing therapy over the contralateral of the points reported as the three most painful points in the McGill-Melzack Pain Scale (virtual painful points) to this group in a virtual reality environment
  Interventions: Other: Breathing exercise

INTERVENTIONS:
Other: Breathing exercise — Breathing exercises will include;
  1. Correct posture and sitting
  2. Nose opening techniques
  3. Diaphragmatic breathing, which consists of continuous and deep nasal inspiration with movement of the abdominal region and diaphragm
  4. Main Breathing exercise (during 5 minutes)=inspiration (during 5 seconds) + expiration (during 15 seconds).

SUMMARY:
Fibromyalgia (FM) is a chronic pain syndrome characterized by impaired perception, transmission, and processing of nociceptive stimuli and causing widespread pain. Pain in FM is the disease itself and is characterized by nociplastic pain that may occur independently of any peripheral nociceptor activity or be felt without disease or damage to the somatosensory system. It is thought that the pain processing process is disrupted due to the changing neurotransmitter release activity and this situation causes pain to be felt more in FM. Chronic pain is the result of perception alteration associated with nociceptive afferent information affecting the cortex; underlying this change are limbic emotional learning mechanisms. Numerous factors, including emotional state, attention, and past painful experiences, modulate nociceptive inputs with the activation of multiple brain regions, resulting in a personalized pain experience. The chronic pain management program should target the central nervous system rather than the peripheral tissues because pain originates in the sensitized nervous system. For this reason, it is important to include plasticity-oriented approaches, cortical disinhibition methods, and strategies for improving perception and behavior change, which aim to replace negative beliefs with positive beliefs, into clinical practice. Our project aims to investigate the effectiveness of the therapeutic intervention, which consists of patient education supported Neuro-Linguistic Programming (NLP), visual feedback and metaphor-assisted breathing therapy designed to provide a perception of improvement and presented in a virtual reality environment, on pain processing, pain intensity, pain-pressure threshold, psychosomatic reflections (biomechanical and viscoelastic properties of tissue, sleep quality, pain catastrophizing behavior, anxiety and depression), disease impact and quality of life in FM patients.

ELIGIBILITY:
Inclusion Criteria:

Diagnosed with Fibromyalgia at least 1 year ago according to ACR criteria

Age range 25-55

Female

Scored at least 24 on the Mini-Mental State Assessment Test

Reported weekly pain intensity of at least 40 mm on the Visual Analog Scale

Be on a stable dose of medication for at least 6 months (serotonin norepinephrine reuptake inhibitors [e.g., duloxetine, milnacipran]; alpha 2-delta receptor ligand [e.g., pregabalin]; gabapentinoids)

Exclusion Criteria:

Having inflammatory rheumatic disease, malignancy, neurological disease, connective tissue disease, severe anemia, uncontrolled endocrine diseases

Body Mass Index (BMI) ≥ 30 Kg/m2

Being pregnant

Having inability to understand, read and speak Turkish

Having difficulty in hearing and seeing

Having any metallic or electronic device in the body that will create incompatibility with the magnetic field in the fMRI scan Having any disease diagnosis (serious psychotic disorder, delirium, mental retardation, epilepsy, heart disease, lung diseases, etc.) that may prevent participation in the evaluation and training to be conducted within the scope of the research

Ages: 25 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Fibromyalgia patient
Enrollment: 39 (Estimated)
Dates: Start 2024-08-13 (Actual); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-08-15 (Estimated)

PRIMARY OUTCOMES:
Functional Magnetic Resonance | Measurement of changes from baseline process of processing pain will be measured at 6 week and 10 week
  The process of processing pain will be determined by functional magnetic resonance imaging performed immediately before and after the experimental pressure pain. ROI analysis will ve performed. No score is defined.
Measurement of pain-pressure threshold | Measurement of changes from baseline of pain-pressure threshold will be measured at 6 week and 10 week
  Pain-pressure threshold evaluated with a pain threshold measuring device (Algometer).

SECONDARY OUTCOMES:
Sleep Quality | Measurement of changes from baseline of sleep quality will be measured at 6 week and 10 week
  Sleep quality will be evaluated with Pittsburgh Sleep Quality Index. Score is between 0 (the best sleep quality) and 21 (the worst sleep quality)
Functional status and disease impact | Measurement of changes from baseline of functional status and disease impact will be measured at 6 week and 10 week.
  Functional status and disease impact will be evaluated with Revised Fibromyalgia Impact Questionnaire. Score is between 0 (no disease impact and 100 (the highest disease impact)
Quality of Life of patients | Measurement of changes from baseline of quality of life will be measured at 6 week and 10 week
  Quality of Life will be measured with QOL Short Form 12. Score is between 0 (the lowest quality of life and 100 (the highest quality of life)
Anxiety and Depression Status | Measurement of changes from baseline of anxiety and depression status will be measured at 6 week and 10 week
  Anxiety and Depression will be evaluated with Hospital Anxiety and Depression Scale. Score is between 0 (no anxiety and depression risk) and 21 (the highest anxiety and depression risk)
Pain catastrophizing behavior | Measurement of changes from baseline of changes from baseline of pain catastrophizing behaviors will be measured at 6 week and 10 week
  Assessing pain catastrophizing behavior will be evaluated with Pain Catastrophizing Scale. Score is between 0 (no pain catastrophizing behavior) and 52 (the highest pain catastrophizing behavior)
Patient satisfaction | Measurement of changes from baseline of patient satisfaction will be measured at 6 week and 10 week
  Patient satisfaction will be evaluated with Global Rating of Change. No score is defined.
Measurement of biomechanical characteristics of tissue | Measurement of changes from baseline stiffness values of tissue will be measured at 6 week and 10 week]
  Stiffness values of tissue will be measured with myotonPro B1 over the three most painful points in Control Group and Virtual Reality-1 Group.
  Stiffness values of tissue will be measured with myotonPro B1 over the contralateral of the points reported as the three most painful points in Virtual Reality-2 Group.
Measurement of biomechanical characteristics of tissue | Measurement of changes from baseline tone values of tissue will be measured at 6 week and 10 week]
  Tone values of tissue will be measured with myotonPro B1 over the three most painful points in Control Group and Virtual Reality-1 Group.
  Tone values of tissue will be measured with myotonPro B1 over the contralateral of the points reported as the three most painful points in Virtual Reality-2 Group.
Measurement of biomechanical characteristics of tissue | Measurement of changes from baseline decrement values of tissue will be measured at 6 week and 10 week]
  Decrement values of tissue will be measured with myotonPro B1 over the three most painful points in Control Group and Virtual Reality-1 Group.
  Decrement values of tissue will be measured with myotonPro B1 over the contralateral of the points reported as the three most painful points in Virtual Reality-2 Group.
Measurement of viscoelastic characteristics of tissue | Measurement of changes from baseline creep values of tissue will be measured at 6 week and 10 week]
  Creep values of tissue will be measured with myotonPro B1 over the three most painful points in Control Group and Virtual Reality-1 Group.
  Creep values of tissue will be measured with myotonPro B1 over the contralateral of the points reported as the three most painful points in Virtual Reality-2 Group.
Measurement of viscoelastic characteristics of tissue | Measurement of changes from baseline relaxation time values of tissue will be measured at 6 week and 10 week]
  Relaxation time values of tissue will be measured with myotonPro B1 over the three most painful points in Control Group and Virtual Reality-1 Group.
  Relaxation time values of tissue will be measured with myotonPro B1 over the contralateral of the points reported as the three most painful points in Virtual Reality-2 Group.

CONTACTS AND LOCATIONS:
Overall Officials: Nilüfer Kablan, PhD, Principal Investigator — İstanbul Medeniyet Üniversitesi
Locations (1):
- Nilüfer kablan, Istanbul, Kartal, Turkey (Türkiye)

REFERENCES:
- [Result] Adams LM, Turk DC. Psychosocial factors and central sensitivity syndromes. Curr Rheumatol Rev. 2015;11(2):96-108. doi: 10.2174/1573397111666150619095330. PMID 26088211
- [Result] Arnold LM, Bennett RM, Crofford LJ, Dean LE, Clauw DJ, Goldenberg DL, Fitzcharles MA, Paiva ES, Staud R, Sarzi-Puttini P, Buskila D, Macfarlane GJ. AAPT Diagnostic Criteria for Fibromyalgia. J Pain. 2019 Jun;20(6):611-628. doi: 10.1016/j.jpain.2018.10.008. Epub 2018 Nov 16. PMID 30453109
- [Result] Caneiro JP, Bunzli S, O'Sullivan P. Beliefs about the body and pain: the critical role in musculoskeletal pain management. Braz J Phys Ther. 2021 Jan-Feb;25(1):17-29. doi: 10.1016/j.bjpt.2020.06.003. Epub 2020 Jun 20. PMID 32616375
- [Result] Ciaramella A. Hypnotic analgesia in chronic pain: role of psychopathology and alexithymia. Am J Clin Hypn. 2023 Apr;65(4):299-313. doi: 10.1080/00029157.2022.2161868. Epub 2023 Feb 7. PMID 36749869
- [Result] de la Coba P, Montoro CI, Reyes Del Paso GA, Galvez-Sanchez CM. Algometry for the assessment of central sensitisation to pain in fibromyalgia patients: a systematic review. Ann Med. 2022 Dec;54(1):1403-1422. doi: 10.1080/07853890.2022.2075560. PMID 35579545
- [Result] Gholamrezaei A, Van Diest I, Aziz Q, Vlaeyen JWS, Van Oudenhove L. Controlled breathing and pain: Respiratory rate and inspiratory loading modulate cardiovascular autonomic responses, but not pain. Psychophysiology. 2021 Oct;58(10):e13895. doi: 10.1111/psyp.13895. Epub 2021 Jul 6. PMID 34231231
- [Result] Ichesco E, Puiu T, Hampson JP, Kairys AE, Clauw DJ, Harte SE, Peltier SJ, Harris RE, Schmidt-Wilcke T. Altered fMRI resting-state connectivity in individuals with fibromyalgia on acute pain stimulation. Eur J Pain. 2016 Aug;20(7):1079-89. doi: 10.1002/ejp.832. Epub 2016 Jan 15. PMID 26773435